CLINICAL TRIAL: NCT01817725
Title: Effect of Hepatitis B Vaccine in Chronic Hepatitis B Patients With Low Serum HBsAg-a Pilot Study
Brief Title: Hepatitis B Vaccine in Chronic Hepatitis B Patients With Low Serum HBsAg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Wei Lai, M.D., Ph.D., Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChangGungMH 101-3594A3
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis B
Keywords: Therapeutic vaccine; HBsAg clearance; Immune clearance; HBsAg clearance induced by vaccination; s seroconversion in carriers after vaccination
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Engerix-B (Experimental): Engerix-B (20 μg/ml, GlaxoSmithKline) was administered at 0-2-4-6-8-10-12 months in dosage of 40μg for >20 years old and 20μg for < or =20 years old
  Interventions: Biological: HBV vaccine (Engerix B)

INTERVENTIONS:
Biological: HBV vaccine (Engerix B) — Engerix-B (20μg/ml, GlaxoSmithKline Biologicals) is administered intramuscularly at 0, 2, 4, 6, 8, 10, 12 months. The dosage will be 20μg in those <= 20 years old and 40μg in those > 20 years old.

SUMMARY:
Background:

The HBsAg clearance rate in interferon-treated responders is significantly higher than that in lamivudine-treated responders, implying immune control is the key to HBsAg clearance. There is a good chance to further increase the cure rate if the investigators can enhance the HBV-specific immune response when the HBsAg level already comes to a low level.

Hypothesis: HBsAg-based vaccine can enhance HBsAg clearance in chronic hepatitis B patients whose HBsAg already <=2000 IU/ml.

Patients and methods:

This pilot study will enroll 20 chronic hepatitis B patients with HBsAg ≦2000 IU/ml, no hepatic decompensation, no HIV coinfection, nor clinical immunodeficiency. Engerix-B vaccine (20μg for <20 years old and 40 μg for ≥ 20 years old) will be given every 2 months for one year. HBsAg quantification, anti-HBs, and HBV DNA will be surveyed regularly before each dose during the treatment period and every 3 months for another year following the last dose. Viral and cellular factors will be studied to discover determinants affecting HBsAg clearance.

Aims

1. To elucidate whether HBsAg-based vaccine can reactivate host immunity to eliminate chronic HBV infection in patients with low titer HBsAg.
2. To delineate the doses to response (HBsAg clearance or decline rate) correlation so as to design a feasible schedule for future clinical trials in a larger group of patients.
3. To discover viral and host factors which can be used as biomarkers for personalized vaccine therapy.

DETAILED DESCRIPTION:
Vaccination schedule:

Engerix-B (20μg/ml, GlaxoSmithKline Biologicals) will be administered intramuscularly at 0, 2, 4, 6, 8, 10, 12 months or until HBsAg clearance. The dosage will be 20μg in those <= 20 years old and 40μg in those > 20 years old.

HBsAg and anti-HBs:

qHBsAg will be checked by commercial kits (Elecsys, Roche Diagnostics, Indianapolis, IN) at baseline, right before every dose, and every 3 months following the last dose for one year. ALT, AST, Alpha-fetoprotein, bilirubin and anti-HBs will be checked simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Naïve or treated chronic hepatitis B patients with positive HBsAg and negative HBeAg;
2. Quantitative serum HBsAg (qHBsAg) <2000 IU/ml;
3. No HIV co-infection;
4. No obvious immunodeficiency (such as renal failure, chemotherapy, radiotherapy, immunosuppressant);
5. Aged 3 to 80 years;

Exclusion Criteria:

1. Pregnancy
2. Allergic to HBV vaccine or yeast.
3. Hepatic decompensation

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Wei Lai, Principal Investigator — Chang Gung Memorial Hospital; Chao-Wei Hsu, Principal Investigator — Chang Gung Memorial Hospital; Chau-Ting Yeh, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan Xian, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai MW, Hsu CW, Lin CL, Chien RN, Lin WR, Chang CS, Liang KH, Yeh CT. Multiple doses of hepatitis B recombinant vaccine for chronic hepatitis B patients with low surface antigen levels: a pilot study. Hepatol Int. 2018 Sep;12(5):456-464. doi: 10.1007/s12072-018-9890-x. Epub 2018 Aug 7. PMID 30088198

RESULTS

PARTICIPANT FLOW:
Groups:
- Engerix-B: Engerix-B (20 μg/ml, GlaxoSmithKline) was administered at 0-2-4-6-8-10-12 months in dosage of 40μg for >20 years old and 20μg for < or =20 years old
  HBV vaccine (Engerix B): Engerix-B (20μg/ml, GlaxoSmithKline Biologicals) is administered intramuscularly at 0, 2, 4, 6, 8, 10, 12 months. The dosage is 20μg in those <= 20 years old and 40μg in those > 20 years old.
Period: Overall Study
Arm/Group | Engerix-B
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Engerix-B
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  Taiwan | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in HBsAg Levels From Baseline to 2 Years
Description: The difference of HBsAg levels at the end of follow up (2 years) and baseline
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: log IU/ml
Arm/Group | Engerix-B
Number analyzed (Participants) | 19
log IU/ml | -0.27 (0.48)
Statistical Analysis 1: Comparison: Engerix-B; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Anti-HBs Seropositivity
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B
Number analyzed (Participants) | 19
Participants | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Engerix-B
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This is a pilot study. A control arm is not included. However, from literature review, natural HBsAg decay without seroconversion was around 0.054~0.058 log IU/ml/year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No